CLINICAL TRIAL: NCT00532402
Title: Continuous and Discontinuous Determination of Propofol Concentration in Breathing Gas - Compared With Propofol Concentration in Plasma (Before and) After Lung Passage and Neurophysiological Parameters
Brief Title: Continuous and Discontinuous Determination of Propofol Concentration in Breathing Gas
Status: Completed | Type: Observational
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Martin Grossherr, Consultant, University of Luebeck
Other Study IDs: P-A-S-1
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: General Anesthesia
Keywords: Monitoring; Breathing Gas; Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study should compare the propofol concentration in breathing gas and in plasma (before and) after lung passage. Propofol concentrations in breathing gas are continuously measured by a sensor. For comparison a discontinuous method is used. Neurophysiologic parameters for determination of depth of anesthesia are compared to the continuous measured propofol concentration in breathing gas.

Study hypothesis: continuous measured propofol concentration in breathing gas correlates to propofol concentration in plasma and depth of anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patient destined for general anesthesia

Exclusion Criteria:

* Heart insufficiency NYHA IV
* Allergy to propofol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having general anesthesia for cardiac and non-cardiac operation
Sampling Method: Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2007-09; Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Gehring, MD, PhD, Study Director — Dept of Anesthesiology, UK-SH, Campus Luebeck
Locations (2):
- Germany (2):
  - Dept. of Anesthesiology , UK-SH, Campus Luebeck, Lübeck, Schleswig-Holstein
  - Dept. of Anesthesiology, UK-SH, Campus Luebeck, Lübeck, Schleswig-Holstein

REFERENCES:
- [Result] Grossherr M, Hengstenberg A, Meier T, Dibbelt L, Gerlach K, Gehring H. Discontinuous monitoring of propofol concentrations in expired alveolar gas and in arterial and venous plasma during artificial ventilation. Anesthesiology. 2006 Apr;104(4):786-90. doi: 10.1097/00000542-200604000-00024. PMID 16571975